CLINICAL TRIAL: NCT01544140
Title: A Phase I, Open-label, Single-center Study to Assess the Pharmacokinetics of Midazolam, a CYP3A4 Substrate, in Healthy Subjects When Administered Alone and in Combination With a Single Dose of 800-mg Vandetanib (CAPRELSA)
Brief Title: Study in Healthy Volunteers to Assess the Pharmacokinetics of Midazolam Administered Alone and in Combination With Vandetanib
Acronym: Vandetanib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D4200C00103
Record Dates: First submitted 2012-02-23; First posted 2012-03-05 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Volunteers
Keywords: Phase 1; healthy volunteers; pharmacokinetics; vandetanib; midazolam
MeSH Terms: interventions — Midazolam; vandetanib

ARMS (1):
- midazolam then midazolam + vandetanib (Experimental): Midazolam alone followed by midazolam in combination with vandetanib
  Interventions: Drug: Midazolam; Drug: vandetanib

INTERVENTIONS:
Drug: Midazolam — Oral syrup 7.5 mg, single dose
Drug: vandetanib — Oral tablets, 800 mg, single dose

SUMMARY:
The purpose of this study in healthy volunteers is to assess the Pharmacokinetics (PK) of Midazolam administered alone and in combination with Vandetanib.

DETAILED DESCRIPTION:
A Phase I, Open-label, Single-center Study to Assess the Pharmacokinetics of Midazolam, a CYP3A4 Substrate, in Healthy Subjects When Administered Alone and in Combination with a Single Dose of 800-mg Vandetanib (CAPRELSA)

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study
* specific procedures:

  * Volunteers must be males or females aged 18 to 50 years and with a weight of at least 50 kg and body mass index (BMI) between 18 and 30 kg/m2, inclusive
  * Females must have a negative pregnancy test at screening and on admission to the study center.
  * Females must not be lactating and must be of non-childbearing potential defined as postmenopausal or documentation of irreversible surgical sterilization.

Exclusion Criteria:

* History of any clinically significant disease or disorder such as gastrointestinal, hepatic, renal or skin disease.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity,
* Volunteers who smoke more than 5 cigarettes per day or are unable to refrain from smoking while resident in the study center
* Screening blood pressure of greater than 140/90 mmHg and/or a resting heart rate of less than 45 beats per minute (repeat test allowed at the Investigator's discretion)
* Clinically significant abnormal12-lead ECG as assessed by the Investigator,
* QTcF interval greater than 450 ms
* Any positive result on screening for:

  * serum hepatitis B surface antigen,
  * hepatitis C antibody, and
  * human immunodeficiency virus (HIV), or
* Positive screen for drugs of abuse.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
AUC for midazolam administered alone and in combination with vandetanib 800 mg | Predose,0.5,1,1.5,2,3,4,6,8,12,16,24,30,36,48 hrs post dose
Cmax for midazolam administered alone and in combination with vandetanib 800 mg | Predose,0.5,1,1.5,2,3,4,6,8,12,16,24,30,36,48 hrs post dose

SECONDARY OUTCOMES:
Frequency and severity of adverse events | Treatment period from 7 to 14 days
ECG data | Treatment period from 7 to 14 days
Laboratory data | Treatment period from 7 to 14 days
Vital signs data | Treatment period from 7 to 14 days
Other PK parameters for midazolam administered alone and in combination with vandetanib 800 mg | Predose,0.5,1,1.5,2,3,4,6,8,12,16,24,30,36,48 hrs post dose
Vandetanib PK parameters for vandetanib in combination with midazolam | Predose,1,2,3,4,5,6,7,8,10,12,18,24,36,48,72,96,120,144,168,192,216 hrs post dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Johansson S, Read J, Oliver S, Steinberg M, Li Y, Lisbon E, Mathews D, Leese PT, Martin P. Pharmacokinetic evaluations of the co-administrations of vandetanib and metformin, digoxin, midazolam, omeprazole or ranitidine. Clin Pharmacokinet. 2014 Sep;53(9):837-47. doi: 10.1007/s40262-014-0161-2. PMID 25117183
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1438&filename=CSR-D4200C00103.pdf
- See also: CSR-D4200C00103.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1438&filename=CSR-D4200C00103.pdf
- See also: Revised_CSP_redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1438&filename=D4200C00103_Revised_CSP_redacted.pdf